CLINICAL TRIAL: NCT00087269
Title: Phase II Study to Evaluate the Tumor Biochemical Effects of the EGFR Tyrosine Kinase Inhibitor OSI-774 (Erlotinib) Administered Prior to Surgical Resection in Patients With Early Stage Non-Small Cell Lung Cancer
Brief Title: Erlotinib in Treating Patients With Stage I-IIIA Non-Small Cell Lung Cancer Undergoing Surgical Resection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02950; E4503; U10CA021115 (NIH)
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Stage IA Non-small Cell Lung Cancer; Stage IB Non-small Cell Lung Cancer; Stage IIA Non-small Cell Lung Cancer; Stage IIB Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

ARMS (1):
- Treatment (erlotinib) (Experimental): Patients receive oral erlotinib once daily on days 1-14 or days 1-21 in the absence of unacceptable toxicity. Patients then undergo surgical resection on the last day of study drug administration (day 14 or day 21). Patients may receive chemotherapy and/or radiotherapy after surgical resection at the discretion of the primary physician.
  Interventions: Drug: erlotinib hydrochloride; Procedure: therapeutic endoscopic surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Procedure: therapeutic endoscopic surgery — Undergo surgical resection
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well erlotinib works in treating patients with stage I, stage II, or stage IIIA non-small cell lung cancer. Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Giving erlotinib before surgery may shrink the tumor so that it can be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the biochemical response rate (> 75% decrease in P-MAPK and/or P-AKT) with daily oral OSI-774 (erlotinib) for 14 consecutive days in patients with early stage, operable NSCLC.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerance of daily oral OSI-774 (erlotinib) as pre-operative treatment for early stage operable NSCLC.

TERTIARY OBJECTIVES:

I. To correlate antiproliferative (Ki-67, p27) and apoptotic (TUNEL assay) tumor responses to OSI-774 (erlotinib) with pre-therapy tumor and skin EGFR pathway functional status and post-therapy tumor and skin EGFR pathway inhibition in patients with resectable NSCLC treated preoperatively with OSI-774 (erlotinib) for 14 days.

II. Assessment of functional EGFR status: HER1, HER-2, HER3, HER4, PHER1, AKT, P-AKT, MAPK-P-MAPK, STAT-3, P-STAT-3, EGFR-III by immunohistochemistry (IHC).

III. Assessment of proliferative response: Ki67 and p27 by IHC. IV. Assessment of apoptotic response: TUNEL assay. V. To study the role of the gastrin-releasing factor and estrogen receptor pathways in the sensitivity and resistance of NSCLC to OSI-774 (erlotinib).

VI. To identify patterns of gene and protein expression pre-therapy and post-therapy that are associated with tumor clinical, biochemical, antiproliferative, and apoptotic responses.

VII. To study the antitumor activity of OSI-774 (erlotinib) in NSCLC tumors heterotransplanted in nude mice after surgical resection and to investigate the sequential molecular changes associated with tumor response to OSI-774 (erlotinib) therapy.

OUTLINE: This is a multicenter study.

Patients receive oral erlotinib once daily on days 1-14 or days 1-21 in the absence of unacceptable toxicity. Patients then undergo surgical resection on the last day of study drug administration (day 14 or day 21). Patients may receive chemotherapy and/or radiotherapy after surgical resection at the discretion of the primary physician.

Patients are followed for 5 years after study registration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspicion of lung cancer without distant metastases
* Patients are scheduled to have a tissue diagnostic procedure within 3 to 5 days of pre-registration
* Patients are willing to allow collection and submission of baseline and post-therapy tumor tissue, skin and blood samples for this study
* Patients must have ECOG performance status of 0, 1, or 2
* Patients must have no psychological, familial, sociological, or geographic conditions that will interfere with medical follow-up and compliance with the study protocol
* Patients must have no prior chemotherapy or radiation therapy or no prior anti- EGFR treatment exposure
* Patients must be able to take oral medication and not have malabsorption syndrome, or prior gastrointestinal surgery that limits their absorption (i.e. requiring total parental nutrition)
* Patients must not be using phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital, oxcarbazepine, rifapentine, St John's Wort, or any other CYP 3A4 enzyme-inducing agent; any use of these substances must be discontinued at least 2 weeks prior to registration
* Patients must not be taking any anti-coagulants
* Patients must not have been treated with a non-approved or investigational drug within 21 days prior to pre-registration; patients must not have serious underlying medical condition that would impair the ability of patient to receive the planned treatment
* Patients with a known hypersensitivity to OSI-774 (erlotinib) are not eligible
* Patients must have histologically confirmed NSCLC; cytologic specimens obtained by brushing, washing or needle aspiration of defined lesions will be acceptable
* Patients must have stage IA (T1N0M0), stage IB (T2N0M0), stage IIA (T1N1M0), stage IIB (T2N1M0; T3N0-1M0), or stage IIIA (T1-3N2M0) disease
* Patients with small cell component on histology specimen are not eligible
* A paraffin-embedded cell block and 1-2 segments of frozen tissue demonstrating NSCLC and obtained during the diagnostic biopsy is available for submission
* Patients must be considered operable candidates and disease must be considered resectable
* Pregnant or breastfeeding women are excluded from the study because the agents used in this study may be teratogenic to a fetus or child and there is no information on the excretion of the agents or their metabolites into breast milk

  * All females of childbearing potential must have a blood test or urine study within 1 week, prior to registration to rule out pregnancy
  * Women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of contraception
* WBC >= 3500/mm^3
* ANC >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Total bilirubin < 1.5mg/dL
* SGPT and SGOT < 3 times institution's upper limit of normal
* Serum creatinine < 2mg/dl or creatinine clearance >= 20 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2004-12; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Biochemical response rate in tumor defined as > 75% decrease in P-MAPK and/or P-AKT | Up to 5 years

SECONDARY OUTCOMES:
Tolerability of erlotinib, graded according to the NCI CTCAE version 3.0 | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Keller, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States